CLINICAL TRIAL: NCT05126810
Title: Evaluate Willingness to Participate in a Trial Comparing Standard Genetic Counseling Versus Personalized Genetic Counseling Based on LFSPRO-ShinyApp Data
Brief Title: Willingness to Participate in a Trial Comparing Standard Genetic Counseling Versus Personalized Genetic Counseling
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2021-0151; NCI-2021-10716 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2021-0151 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-10-25; First posted 2021-11-19 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Li-Fraumeni Syndrome
MeSH Terms: conditions — Li-Fraumeni Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Observational (questionnaire): Patients complete a questionnaire over 15-20 minutes. Patients positive for a TP53 mutation complete an additional questionnaire over 15-20 minutes within 1 month after test results.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Other: Questionnaire Administration — Complete questionnaire

SUMMARY:
This study evaluates patients willingness to participate in a trial comparing standard genetic counseling versus personalized genetic counseling. Collecting information from patients may help researchers learn why patients may or may not take part in the future study that compares standard genetic counseling to personalized genetic counseling.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate patients' willingness to participate in a future randomized trial comparing standard genetic counseling versus personalized genetic counseling based on Li-Fraumeni syndrome patient reported outcome (LFSPRO) ShinyApp data.

OUTLINE:

Patients complete a questionnaire over 15-20 minutes. Patients positive for a TP53 mutation complete an additional questionnaire over 15-20 minutes within 1 month after test results.

ELIGIBILITY:
Inclusion Criteria:

* Individuals age 15 or older OR parent/guardian of a patient younger than 15 years (if age 15-17, the patient will provide assent and parent/guardian will provide consent), pregnant women will also be allowed to participate
* English fluency
* Receive genetic counseling specifically for TP53 genetic testing and who consent to undergo TP53 genetic testing OR individuals whose genetic testing indicates a TP53 germline mutation

Exclusion Criteria:

* Individuals who are non-English speaking
* Individuals having low suspicion for a TP53 germline mutation during pretest counseling and test negative for a TP53 mutation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Receive receiving genetic counseling specifically for TP53 genetic testing
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-10-02 (Estimated)

PRIMARY OUTCOMES:
Patient willingness to participate in a future randomized trial comparing standard genetic counseling versus personalized genetic counseling based on LFSPRO ShinyApp data | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Banu Arun, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson Cancer Center — http://www.mdanderson.org